CLINICAL TRIAL: NCT05122052
Title: Effect of Gender on Distress and Fatigue Over Time in Cancer Patients. A Prospective Longitudinal Study.
Brief Title: Effect of Gender on Distress and Fatigue in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Director of Medical Oncology, Ente Ospedaliero Ospedali Galliera
Other Study IDs: 028/2019
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: distress; gender; fatigue; time; effect modification
MeSH Terms: conditions — Neoplasms; Coitus; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women with cancer: Patients with cancer of any site and stage defined as feminine both from the biological (female sex) and psychosocial point of view (feminine gender)
  Interventions: Other: Psychological session
- Men with cancer: Patients with cancer of any site and stage defined as masculine both from the biological (male sex) and psychosocial point of view (masculine gender)
  Interventions: Other: Psychological session

INTERVENTIONS:
Other: Psychological session — Just before the oncology visit, each patient is invited to undergo a psychological session of 20-30 minutes. During the session with a psycho-oncologist the following tasks are addressed: 1) favor emotional expression identifying the most difficult issues to promote mechanisms of elaboration of living experiences; 2) offer a containment of intense emotions; 3) assess awareness of diagnosis and prognosis; 4) favor expression of fears of treatment expectancy; 5) favor expression of difficulties on the inability to cope with prior commitments after the disease; 6) assess family and friend network; 7) improve the patient medic communication and relationship. At the end of the session, the distress thermometer and ESAS-r scale are compiled together with the demographic characteristics. All outstanding issues that are relevant to the therapeutic plan are then discussed between the psychotherapist and the medic before the oncology visit together with delivery of the DT and ESASr scale result.

SUMMARY:
Distress in cancer patients has been shown to be higher in females than males, but the behavior of distress during time in longitudinal prospective studies has not been studied, nor is it known if there are differences related to gender during time. These differences may have important therapeutic implications in terms of selective psychological support as cancer progresses during individual trajectories.

The aim of the present study is to examine the effect of gender during time on psychological distress and fatigue in cancer patients across a broad range of cancer types. It is hypothesized that women will report higher psychological distress than men at initial visit but a reversed trend will be observed during follow-up as a result of different coping capabilities between men and women. We will also investigate if psychological factors (distress, anxiety and depression) affected antibody response and markers of COVID-19 vaccine activation (C-reactive protein, CRP and D-dimer) after 6 months from initial vaccination.

Caregivers will also be interviewed to measure their burden with the Zarit Burden Interview.

Patients attending a cancer outpatient clinic are invited to undergo a psychological session immediately before the medical visit. Distress is assessed by the Distress thermometer and fatigue by the ESAS-r scale at the end of the session. Patients will undergo follow-up visits to assess changes during time and possible time by gender interactions.

DETAILED DESCRIPTION:
Distress and fatigue in cancer patients are important factors affecting treatment compliance and efficacy and quality of life. The prevalence of moderate or severe emotional distress in cancer patients ranges from 30 to 45% depending on a point of assessment. The National Comprehensive Cancer Network indicates that all cancer patients should undergo a distress measurement as the sixth vital parameter to prevent more serious psychological disorders, including anxiety, depression and coping disturbances. Several studies indicate that patients undergoing psychotherapy or psychosocial support to relieve cancer distress have better disease coping, a reduction of fatigue, anxiety and depression and an improvement in quality of live and possibly survival.

Distress in cancer patients has been shown to be higher in females than males, but the behavior of distress during time in longitudinal prospective studies has not been studied, nor is it known if there are differences related to gender during time. These differences may have important therapeutic implications in terms of selective psychological support as cancer progresses during individual trajectories.

The aim of the present study is to examine the effect of gender during time on psychological distress and fatigue in cancer patients across a broad range of cancer types. It is hypothesized that women will report higher psychological distress than men at initial visit but a reversed trend will be observed during follow-up as a result of different coping capabilities between men and women.

In a subset of patients, we will also investigate if psychological factors (distress, anxiety and depression) affected antibody response and markers of COVID-19 vaccine activation (C-reactive protein, CRP and D-dimer) after 6 months from initial vaccination.

Caregivers will also be interviewed with the Zarit questionnaire, a popular caregiver self-report measure used by many aging agencies, originated as a 29-item questionnaire The 29-item instrument is included in Zarit et al., 1980. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).

Patients attending a cancer outpatient clinic are invited to undergo a psychological session immediately before the medical visit. Distress is assessed by the Distress thermometer and fatigue by the ESAS-r scale at the end of the session. Patients will undergo follow-up visits to assess changes during time and possible time by gender interactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer of any site and stage willing to undergo a psychological interview before the medical visit, including those receiving COVID-19 vaccine.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Study Population: Patients with cancer of any site and stage willing to undergo a psychological interview before the medical visit.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Cancer distress | 3 years
  The patient rates his/her level of distress over the past week after the psychological session. The Distress Thermometer (DT) was developed as a simple tool to effectively screen for symptoms of distress. The instrument is a self-reported tool using a single-item tool using a 0 (no distress) to 10 (extreme distress)-point Likert scale resembling a thermometer. Additionally, the patient is prompted to identify sources of distress using a 39-item supplemental list of potential sources of distress, including the following domains: emotional, physical, practical, family, and spiritual/religious problems. DT scores are categorized in three levels, 0-3, low, 4-6, moderate, 7-10, severe. The DT has demonstrated adequate reliability and has been translated and validated into numerous languages, including Italian.

SECONDARY OUTCOMES:
Cancer fatigue | 3 years
  The Edmonton Symptom Assessment System (ESAS) represents one of the first symptom batteries in palliative care to support symptom assessment in many centers worldwide. A revised ESAS numeric rating scale (ESAS-r) consisting of 9 core symptoms (pain, tiredness, nausea, depression, anxious, drowsiness, appetite, feeling of well being, shortness of breath) and an optional 10th symptom has more recently been developed. Specifically, ESAS-r stated the time frame of symptom assessment as "now", added brief explanations for tiredness ("lack of energy"), drowsiness ("feeling sleepy"), depression ("feeling sad") and anxiety ("feeling nervous") and well-being ("how you feel overall"), changed "appetite" to "lack of appetite", adjusted the order of symptoms, removed the horizontal line over the numbers and shaded alternate items in gray for readability, and sugge

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Rondanina, PhD, Study Chair — Ente Ospedaliero Ospedali Galliera
Locations (1):
- E.O. Ospedali Galliera, Genova, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication of the trial will be shared (text, tables, figures, and appendices), after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared 3 months following the publication of the article and they will remain available for 36 months.
Access Criteria: The investigators who would like to use the data have to prepare a proposal that needs to be approved the Steering committee. The aim of the access to study data needs to be specified in the proposal. Proposals should be sent to the Principal investigator (andrea.decensi@galliera.it). To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Bultz BD, Carlson LE. Emotional distress: the sixth vital sign--future directions in cancer care. Psychooncology. 2006 Feb;15(2):93-5. doi: 10.1002/pon.1022. No abstract available. PMID 16444764
- [Background] Moro C, Brunelli C, Miccinesi G, Fallai M, Morino P, Piazza M, Labianca R, Ripamonti C. Edmonton symptom assessment scale: Italian validation in two palliative care settings. Support Care Cancer. 2006 Jan;14(1):30-7. doi: 10.1007/s00520-005-0834-3. Epub 2005 Jun 4. PMID 15937688
- [Background] Faller H, Weis J, Koch U, Brahler E, Harter M, Keller M, Schulz H, Wegscheider K, Boehncke A, Hund B, Reuter K, Richard M, Sehner S, Szalai C, Wittchen HU, Mehnert A. Perceived need for psychosocial support depending on emotional distress and mental comorbidity in men and women with cancer. J Psychosom Res. 2016 Feb;81:24-30. doi: 10.1016/j.jpsychores.2015.12.004. Epub 2015 Dec 15. PMID 26800635
- [Background] Boyes A, Newell S, Girgis A, McElduff P, Sanson-Fisher R. Does routine assessment and real-time feedback improve cancer patients' psychosocial well-being? Eur J Cancer Care (Engl). 2006 May;15(2):163-71. doi: 10.1111/j.1365-2354.2005.00633.x. PMID 16643264
- [Background] Rondanina G, Siri G, Marra D, DeCensi A. Effect of sex on psychological distress and fatigue over time in a prospective cohort of cancer survivors. J Cancer Surviv. 2024 Apr;18(2):586-595. doi: 10.1007/s11764-022-01291-z. Epub 2022 Nov 7. PMID 36344904